CLINICAL TRIAL: NCT03442543
Title: A Novel Technique for Preoperative Localization of Sentinel Lymph Node in Breast Cancer Patients by Silver Wire Insertion or Liquid Charcoal Injection Guided by CT Lymphography
Brief Title: Preoperative Localization of Sentinel Lymph Node in Breast Cancer Patients By Novel Computed Tomography-Lymphography Guided Technique
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Omar Hamdy, Principal investigator, Assistant lecturer of surgical oncology, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: MD/17.03.68
Record Dates: First submitted 2018-02-16; First posted 2018-02-22 (Actual); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Breast Cancer
Keywords: sentinel lymph node biopsy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- charcoal (Experimental)
  Interventions: Device: preoperative localization of SLN detected by CTLG by either methods
- silver wire (Experimental)
  Interventions: Device: preoperative localization of SLN detected by CTLG by either methods

INTERVENTIONS:
Device: preoperative localization of SLN detected by CTLG by either methods — 50 patients with node negative early breast cancer. The patients were randomized into two groups; SLN localized using CTLG guided injection of liquid charcoal suspended solution (first group) or by placing a 3 cm silver wire using spinal needle (second group). For every patient, SLN biopsy was performed using the traditional method with blue dye. Then dual search for the SLN localized by both the novel & traditional method was performed.

SUMMARY:
A question is raised about the possibility of accurate localization of the SLN (sentinel lymph node) detected by CTLG (Computed Tomography Lymphography) which offers a detection rate of 100% in many studies In Oncology center, Mansoura University (OCMU), the surgical oncology unit had a previous experience in using charcoal for localization of non-palpable suspicious breast lesions and it showed promising results in comparison to traditional localization methods In addition, we had another study using silver wire for localization of breast masses before neoadjuvant therapy.

In the study, the investigators will study the usage of both methods as preoperative localization methods for the SLN detected by CT lymphography in breast cancer patients The investigators suppose that this method can offer two main advantages over the traditional SLN intraoperative methods which are; saving operative time needed for the intraoperative procedure as well as solving the problem of the need for complex logistic preparations especially for the usage of radioisotope method.

ELIGIBILITY:
Inclusion Criteria:

* node negative early breast cancer

Exclusion Criteria:

* • Unfit patients for general anaesthesia

  * Previous axillary surgery
  * History of breast surgery or incisional biopsy compromising the breast lymphatic drainage.
  * Known hypersensitivity to the dye
  * Patients with clinically positive or suspicious axilla
  * Pregnant females

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-07-02 (Actual); Primary Completion 2018-07-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
detection of the sentinel lymph node by the novel method & matching between the sentinel lymph node detected by the novel method and the control one | one year

CONTACTS AND LOCATIONS:
Overall Officials: Omar Hamdy, MSc, Principal Investigator — Oncology center, Mansoura University
Locations (1):
- Oncology center, Mansoura University, Al Mansurah, Egypt